CLINICAL TRIAL: NCT00518830
Title: Randomized Clinical Trial for the Treatment of Postnatal Depression
Brief Title: Treatment of Postnatal Depression for Low-Income Mothers in Primary Care in Santiago, Chile
Acronym: DPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1040434
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-07

CONDITIONS: Postnatal Depression
Keywords: postnatal depression; primary care; depressed women
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PND-MCI (Experimental): The multi-component intervention involved a psychoeducational group, treatment adherence support, and pharmacotherapy if needed
  Interventions: Other: multi-component intervention
- usual care (Active Comparator): 'Usual care' included all services normally available in the clinics, including antidepressant medication, brief psychotherapeutic interventions or referral for specialty treatment
  Interventions: Other: Usual care

INTERVENTIONS:
Other: multi-component intervention — The PND-MCI included psycho-educational groups, structured pharmacotherapy if needed, and systematic monitoring of clinical progress and treatment compliance
  Arms: PND-MCI
Other: Usual care — included all services normally available in the clinics, including antidepressant medication, brief psychotherapeutic interventions or referral for specialty treatment
  Arms: usual care

SUMMARY:
A randomized clinical trial was carried out at primary care level in Santiago, Chile to investigate a combined treatment for women suffering post-natal depression and preventing the adverse consequences of this illness on infant's growth and development.

DETAILED DESCRIPTION:
Background: We compared the effectiveness of a multi-component intervention with usual care to treat postnatal depression among low-income mothers in primary care clinics in Santiago, Chile.

Methods: Randomised controlled trial. Two hundred and thirty mothers with major depression attending postnatal clinics were randomly allocated to either a multi-component intervention or usual care. The multi-component intervention involved a psychoeducational group, treatment adherence support, and pharmacotherapy if needed. Data were analysed on an intention-to-treat basis. The main outcome measure was the Edinburgh Postnatal Depression Scale (EPDS) at 3 and 6 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Mothers meeting criteria for current DSM-IV major depression were eligible.

Exclusion Criteria:

* who had received any form of treatment for their depression during their current postnatal period,
* those who were pregnant,
* with psychotic symptoms,
* serious suicidal risk,
* history of mania,
* alcohol or drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2004-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
EPDS | 3 and 6 months

SECONDARY OUTCOMES:
four dimensions of the Short Form-36 (SF-36) Questionnaire: mental health; emotional role; social functioning; and vitality(34) and significant clinical improvement. | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Rojas, MD, Principal Investigator — University of Chile

REFERENCES:
- [Derived] Rojas G, Fritsch R, Solis J, Jadresic E, Castillo C, Gonzalez M, Guajardo V, Lewis G, Peters TJ, Araya R. Treatment of postnatal depression in low-income mothers in primary-care clinics in Santiago, Chile: a randomised controlled trial. Lancet. 2007 Nov 10;370(9599):1629-37. doi: 10.1016/S0140-6736(07)61685-7. PMID 17993363